CLINICAL TRIAL: NCT00677586
Title: Simultaneous Versus Staged Resection for Initially Resectable Synchronous Rectal Cancer Liver-limited Metastasis: A Randomized Controlled Trial
Brief Title: Simultaneous Versus Staged Resection for Initially Resectable Synchronous Rectal Cancer Liver-limited Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Deputy director of the department of general surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESONANCE
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Rectal Neoplasm With Metastasis to the Liver
Keywords: rectal neoplasms; liver metastasis; surgery; simultaneous resection; staged resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Rectal cancer patients with synchronous resectable liver metastasis were randomized to simultaneous resection of primary and metastatic lesions or staged resection
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): simultaneous resection of liver metastasis and the rectal primary tumor
  Interventions: Procedure: simultaneous resection of liver metastasis and the rectal primary tumor
- 2 (Active Comparator): staged resection of the liver metastasis and the rectal primary tumor
  Interventions: Procedure: staged resection of liver metastasis and the rectal primary tumor

INTERVENTIONS:
Procedure: simultaneous resection of liver metastasis and the rectal primary tumor — simultaneous resection of liver metastasis and the rectal primary tumor
  Arms: 1
Procedure: staged resection of liver metastasis and the rectal primary tumor — Patients received resection of the rectal tumor. 1 months later received resection of liver metastasis
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of simultaneous liver resections compared to staged hepatectomies of rectal cancer with liver metastasis and to compare the short and long-term survival between the two groups.

DETAILED DESCRIPTION:
The optimal surgical strategy for treatment of patients with resectable synchronous rectal liver metastases remains controversial. To answer whether synchronous rectal cancer liver metastases (SLM) should be resected simultaneously with primary cancer or should be delayed, We conducted a randomized, controlled trial to compare the safety and efficacy of simultaneous versus delayed resection of the rectum and liver. Patients with rectal cancer and resectable SLM were randomly assigned to either simultaneous or delayed resection of the metastases. The primary outcome was the rate of major complications (Clavien-Dindo grade≥III) within 30 days following surgery. Secondary outcomes included disease-free and overall survival. A consecutive patients of rectal cancer with liver metastasis from ZhongShan hospital, Fudan university were enrolled and randomly assigned to simultaneous liver resections and staged hepatectomies. Post-operative complications, peri-operative mortality, long-term survival were compared.

ELIGIBILITY:
Inclusion Criteria:

* age>=18 and <= 75 years
* resectable primary rectal tumor
* remnant liver volume >= 60%
* without other organ metastasis or peritoneum metastasis
* without contradiction of cardiac and pulmonary diseases
* American Society of Anesthesiologists (ASA) class I - II
* Histologically proved rectal adenocarcinoma

Exclusion Criteria:

* age > 75 years
* unresectable primary rectal tumor
* remnant liver volume < 60%
* with other organ metastasis or peritoneum metastasis
* with contradiction of cardiac and pulmonary diseases
* Tumors assessed as clinical complete response after preoperative radio- or chemoradiotherapy
* Signs of acute intestinal obstruction, bleeding or perforation needing emergency surgery
* Multiple colorectal tumors or other schedules needing for synchronous colon surgery
* Co-existent inflammatory bowel disease
* Pregnancy or lactation
* Patients received treatment other than preoperative radio- or chemoradiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Severe complication rate after resection of primary and metastatic lesions | 30 days after surgery
  Grade of III-V complication rate according to Clavien-Dindo

SECONDARY OUTCOMES:
Disease free survival | 3 years
  Disease free survival after the last resection of primary and metastatic lesions
Overall survival | 3 years
  Overall survival after the last resection of primary and metastatic lesions
Post-operative mortality | 90 days after surgery
  any death occured within 90 days after the last resection of primary and metastatic lesions
Cost of hospitalization | 2 months
  any cost during the resection of primary and metastatic lesions
Complication rate after resection of primary and metastatic lesions | 30 days after surgery
  All grade of complication rate according to Clavien-Dindo
Postoperative hospital stay | 30 days after surgery
  The postoperative hospital stay is defined as the number of date from the first day after operation to discharge

CONTACTS AND LOCATIONS:
Overall Officials: jianmin xu, MD, PHD, Study Director — department of general surgery, zhongshan hospital, fudan university